CLINICAL TRIAL: NCT06991803
Title: Effects of Different Irrigation Activation Techniques on the Healing of Large Periapical Lesions: A Prospective Clinical Study
Brief Title: Effects of Different Irrigation Activation Techniques on the Healing of Large Periapical Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Recep Tayyip Erdogan University (Other)
Responsible Party: Principal Investigator, Medine Ciçek, endodontist, Recep Tayyip Erdogan University
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MCiçek
Record Dates: First submitted 2025-05-09; First posted 2025-05-28 (Actual); Results first posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Periapical Periodontitis; Irrigation Activation; Lasers
Keywords: Fractal analysis; Irrigation activation; paı; pıps; sweeps; healing of periapical lesion
MeSH Terms: conditions — Periapical Periodontitis

STUDY DESIGN:
Intervention Model Description: A Prospective Clinical Study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: After the preparation was completed, final irrigation was applied via the determined irrigation method.
  The researchers who conducted the PAI and lesion size evaluations were blinded to the irrigation method and preoperative measurements.
  Fractal analysis (FA) was performed by an experienced oral and maxillofacial radiologist who was blinded to the activation method and used the fractal box counting method on panoramic radiographs with ImageJ.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Control Group (Conventional Syringe Irrigation) (Other): In this group, the traditional syringe method was used for final irrigation of the root canals. The canals were irrigated with 6 mL of 17% EDTA solution, 2 mL of saline and, finally, 6 mL of 2.5% NaOCl, and a 30-gauge perforated irrigation needle placed 1-2 mm shorter than the working length was used. During irrigation, 1-2 mm updown movements were made with a constant low pressure.
  Interventions: Other: root canal treatment and irrigation activation
- Group 1 (MDA) (Experimental): After the root canal was filled with irrigation solution, a gutta-percha cone compatible with the master file was positioned 1 mm behind the working length and moved up and down with 100 strokes/minute for activation.
  Interventions: Other: root canal treatment and irrigation activation
- Group 2 (Sonic Activation) (Experimental): Sonic activation was performed via the Easydo Activator device (EA; Easyinsmile (Weixiaomeichi, Changsha, China). While the solution was present in the canal, the needle tip of the device was placed in the canal 2 mm behind the determined working length, and the solutions were activated at the recommended power setting.
  Interventions: Other: root canal treatment and irrigation activation
- Group 3 (PUI) (Experimental): Solutions were activated via ultrasonic tips (mode:E, setting:6) (DTE, Guilin Woodpecker Co., Guilin, Guangxi, China) and an ultrasonic device (DTE S6 Led, Guilin Woodpecker Co., Guilin, Guangxi, China). An ultrasonic tip one size smaller than the master apical file was used 2 mm behind the working length without contacting the walls.
  Interventions: Other: root canal treatment and irrigation activation
- Group 4 (PIPS) (Experimental): A Fotona Er:YAG laser device (LightWalker Fotona, Ljubljana, Slovenia) was used for activation. A special conical and radial fiber tip (PIPS 300/14, Fotona) was placed in the coronal part of the pulp chamber, and the irrigation solutions in the canal were activated in SSP mode (50 μs, 0.3 W, 15 Hz and 20 mJ) with the air and water settings turned off.
  Interventions: Other: root canal treatment and irrigation activation
- Group 5 (SWEEPS) (Experimental): A Fotona Er:YAG laser device (SWEEPS 600, Fotona) with an 8.5 mm long and 600 µm diameter tapered fiber tip was used for activation. The device was set to SWEEPS mode with two ultrashort micropulses (25 μs) continuously changing at 0.3 W, 20 mJ, and 15 Hz. The tip was placed in the pulp chamber, and the solution was activated with the air and water settings turned off.
  Interventions: Other: root canal treatment and irrigation activation

INTERVENTIONS:
Other: root canal treatment and irrigation activation — After the teeth were isolated with a rubber dam, the endodontic access cavity was opened. Then, #10-15 K-type hand files were inserted into the canals, and after determining point 0.0 with the electronic apex locator, the working length was determined to be 0.5 mm shorter than this point and confirmed radiographically. When a discrepancy was observed, the apex locator was considered correct. The root canals were prepared with ProTaper Next up to 3 sizes larger than the initial diameter via a torque-controlled endodontic motor in 300 rpm/2-5.2 Ncm rotation mode. Between each file, the canals were irrigated with 5 ml of 2.5% NaOCl. In retreatment cases, after opening the access cavity under rubber dam isolation, the guta percha was removed with RT files, and the rest of the procedure was performed in the same manner as for primary root canal treatment.

SUMMARY:
The primary goal of endodontic treatment is to treat the infection by optimally cleaning the root canal system and precentig reinfection. Root canal preparation must be accompanied by an effective irrigation activation protocol to effectively remove foci of infection.

Manual dynamic activation (MDA) is an irrigation activation method performed by up- and downmovements of a gutta-percha compatible with the final instrumentation size.Passive ultrasonic irrigation (PUI) is another activation technique based on the transmission of acoustic energy to the irrigant in the canal through a vibrating file or a thin wire with hydrodynamic activation. Sonic systems create a strong hydrodynamic phenomenon and increase the effectiveness of the solution by using flexible tips connected to special instruments that work with air pressure with low-frequency vibration. Recently, laser activation methods, defined as photon-initiated photoacoustic streaming (PIPS) and shock wave enhanced emission photoacoustic streaming (SWEEPS), which work with conical and radial fiber tips, have been developed. The main difference between PIPS and SWEEPS is that in SWEEPS, the double laser pulse applied to the irrigation solution causes the bubbles to collapse faster, allowing the photoacoustic shock wave to reach deeper into the root canal.

Apical periodontitis is a condition in which microbial products in the root canal reach the periapical region, destroy adjacent bone tissue, and is characterized by a radiolucent area in the periradicular region of the affected tooth on a radiograph. Successful healing of apical periodontitis requires a reduction in the size of the radiolucent area and healing of the bone. The periapical index (PAI) system, which grades periapical pathology from 1 to 5 according to increasing radiographic appearance, helps to achieve consensus among clinicians in categorizing lesions. In addition, the healing process of chronic apical periodontitis can be objectively examined via fractal analysis, which can be used to assess the size and density of periapical lesions, the degree of healing of bone tissue, and the remodeling of the trabecular structure quantitatively.

The aim of this study was to compare the effects of different irrigation activation methods (MDA, Sonic, PUI, PIPS, and SWEEPS) on healing in single-rooted mandibular premolar teeth with extensive periapical lesions of endodontic origin.

DETAILED DESCRIPTION:
MATERIALS AND METHODS Local ethics committee approval was obtained from the Recep Tayyip Erdoğan University Ethical Committee (No: 2023/136). All the participants were informed about the study protocol, and written informed consent was obtained.

Sample size calculation The G Power 3.1.9.4 (University Kiel, Germany) program was used to calculate the effect size. The effect size was calculated on the basis of the data of Verma et al., who compared the success of different irrigation techniques in healing after one year. On the basis of the chi-square test data, an effect size of 0.388 was found to be sufficient for significance, and it was calculated that a total of at least 110 samples were required with a type 1 error of 0.05 and 90% power.

Patient selection Vertucci Class I single-rooted mandibular premolars with asymptomatic apical periodontitis and a periapical index (PAI) score of 3 or higher were included in the study. Patients with systemic diseases, bone metabolism diseases and/or drugs that affect bone metabolism (steroids and bisphosphonates) were excluded from the study. Immunocompromised patients, patients with a history of radiotherapy, pregnant patients, teeth with Miller 2 or more mobility, teeth with a periodontal pocket depth of ≥5 mm, teeth with internal and external resorption, and teeth with vertical and horizontal root fractures were excluded. Out of 150 patients aged 18 years and over, a total of 18 patients who refused to participate or did not meet the inclusion criteria were excluded from the study, and 132 patients were included. Pretreatment panoramic radiographs were obtained with a Planmeca Promax 2D S2 device (Planmeca Romexis, Helsinki, Finland). The patients were positioned so that the sagittal plane was parallel to the vertical plane of the dental panoramic machine and the Frankfurt plane was parallel to the floor. The same radiographic exposure settings (66 kVp, 8 mA and 16.6 second exposure time) were used for all patients. For each tooth, the vertical, horizontal and diagonal dimensions passing through the center of the lesion were measured via ImageJ v1.52 software (National Institutes of Health, Bethesda, United States), and the largest dimension obtained was recorded as the preoperative lesion diameter.

Clinical Procedure After the teeth were isolated with a rubber dam, the endodontic access cavity was opened with a sterile diamond rond bur under water cooling. Then, #10-15 K-type hand files (Dentsply Maillefer, Ballaigues, Switzerland) were inserted into the canals, and after determining point 0.0 with the Root ZX mini electronic apex locator (J. Morita Co., Tokyo, Japan), the working length was determined to be 0.5 mm shorter than this point and confirmed radiographically. When a discrepancy was observed, the apex locator was considered correct. After the initial apical diameter with the largest K-type file trapped in the working length was determined, the root canals were prepared with ProTaper Next (PTN; Dentsply Maillefer, Ballaigues, Switzerland) up to 3 sizes larger than the initial diameter via a torque-controlled endodontic motor (SybronEndo, Glendora, CA, USA) in 300 rpm/2-5.2 Ncm rotation mode. Between each file, the canals were irrigated with 5 ml of 2.5% NaOCl. In retreatment cases, after opening the access cavity under rubber dam isolation, the guta percha was removed with RT files (EndoArt RT, İnci Dental, Turkey), and the rest of the procedure was performed in the same manner as for primary root canal treatment.

After the preparation was completed, final irrigation was applied via the determined irrigation method.

Control Group (Conventional Syringe Irrigation) In this group, the traditional syringe method was used for final irrigation of the root canals. The canals were irrigated with 6 mL of 17% EDTA solution, 2 mL of saline and, finally, 6 mL of 2.5% NaOCl, and a 30-gauge perforated irrigation needle placed 1-2 mm shorter than the working length was used. During irrigation, 1-2 mm updown movements were made with a constant low pressure.

Group 1 (MDA) After the root canal was filled with irrigation solution, a gutta-percha cone compatible with the master file was positioned 1 mm behind the working length and moved up and down with 100 strokes/minute for activation.

Group 2 (Sonic Activation) Sonic activation was performed via the Easydo Activator device (EA; Easyinsmile (Weixiaomeichi, Changsha, China). While the solution was present in the canal, the needle tip of the device was placed in the canal 2 mm behind the determined working length, and the solutions were activated at the recommended power setting.

Group 3 (PUI) Solutions were activated via ultrasonic tips (mode:E, setting:6) (DTE, Guilin Woodpecker Co., Guilin, Guangxi, China) and an ultrasonic device (DTE S6 Led, Guilin Woodpecker Co., Guilin, Guangxi, China). An ultrasonic tip one size smaller than the master apical file was used 2 mm behind the working length without contacting the walls.

Group 4 (PIPS) A Fotona Er:YAG laser device (LightWalker Fotona, Ljubljana, Slovenia) was used for activation. A special conical and radial fiber tip (PIPS 300/14, Fotona) was placed in the coronal part of the pulp chamber, and the irrigation solutions in the canal were activated in SSP mode (50 μs, 0.3 W, 15 Hz and 20 mJ) with the air and water settings turned off.

Group 5 (AutoSWEEPS) A Fotona Er:YAG laser device (SWEEPS 600, Fotona) with an 8.5 mm long and 600 µm diameter tapered fiber tip was used for activation. The device was set to AutoSWEEPS mode with two ultrashort micropulses (25 μs) continuously changing at 0.3 W, 20 mJ, and 15 Hz. The tip was placed in the pulp chamber, and the solution was activated with the air and water settings turned off.

In all the activation groups, 2 mL of 17% EDTA solution (SAVER, Prime Dental, Turkey) was activated for 20 s, and this process was repeated 3 times for a total of 6 mL of EDTA activation in 1 min. Then, 2 mL of saline was applied to the canals for 20 s to prevent the chemical interaction of NaOCl and EDTA. Afterward, 2 mL of 2.5% NaOCl solution (MICROVEM, Turkey) was activated for 20 s, and this procedure was repeated 3 times for a total of 6 mL of NaOCl solution activation in 1 minute.

After the final irrigation, the canals were dried with paperpoint (DiaDent, Heungdeok-gu, Korea) and obturated via the cold lateral compaction method via an ADSeal (Meta Biomed, Cheongju, South Korea) sealer and gutta-percha. The gutta-percha was cut 1 mm below the cemento-enamel junction, and coronal restoration was performed with composite resin (Llis, FGM, Joinville, Brazil). All procedures were performed by a single operator (M.Ç.).

Healing evaluation PAI score and lesion diameter At the 12-month follow-up, panoramic radiographs were taken using the same settings as those used for pretreatment radiography. PAI scores of the treated teeth were recorded, and patients were classified as "healed" (PAI <3) or "unhealed" (PAI ≥3). PAI scoring was performed by 2 endodontists, and in cases of disagreement, a consensus was reached by discussion. Additionally, the widest diameter of the lesion at the follow-up session was measured by an endodontist (M.Ç.) The same method was used for the preoperative measurements. The researchers who conducted the PAI and lesion size evaluations were blinded to the irrigation method and preoperative measurements.

Fractal analysis Fractal analysis (FA) was performed by an experienced oral and maxillofacial radiologist (D.N.G.) who was blinded to the activation method and used the fractal box counting method on panoramic radiographs with ImageJ. The program was downloaded from the internet at https://imagej.nih.gov/ij/download.html. To standardize the size and location of the ROI, a parallel line forming a right angle to the apical and long axes of the tooth was placed 1 mm apical to the root apex (Figure 2). The sequence of steps followed when FD analysis was performed was as follows (Figure 3): All digital images were opened in ImageJ v. 1.52 software (National Institutes of Health), and 30x30 pixel sections were taken from the determined regions and saved in 'tif' format. After the area of interest to be analyzed was cropped, it was saved in 8-bit format and copied. A Gaussian filter (sigma= 35 pixels) was applied to the duplicated image. The blurred image was subtracted from the original image via subtraction. A value of 128 was added to each pixel location, and 128 was set as the threshold value regardless of the initial brightness of the image. The 128 brightness threshold image was converted to binary format. An erosion and dilatation process was applied. The inverted image was skeletonized, and FD analysis was applied to the skeletonized image via the 'box-counting' function.

To assess intraobserver reliability, the lesion diameter and fractal measurements were conducted twice with 2-week intervals by the same researchers in 20% of the teeth involved in the study.

Statistical analysis The Jamovi 2.3.28 statistical program was used for statistical analysis. Normal distribution in the comparisons was evaluated by the Shapiro-Wilk test, Kolmogorov-Smirnov test, Anderson-Darling test and Q-Q graph. Homogeneity between variances was analyzed by Levene's test. Since sex data were categorical, the differences between the groups were analyzed via the chi-square test. Since the distribution of age between groups was found to be normal, it was analyzed by Welch's one-way ANOVA test.

Although a normal distribution was obtained in fractal analysis, Welch's one-way ANOVA test was preferred for the comparison of irrigation groups because the variances were not homogeneously distributed, and pairwise comparisons were made with the Games-Howell test. Before and after comparisons within each group, paired sample t tests were used.

Since a normal distribution could not be obtained, the Kruskal-Wallis test was preferred for the comparison of irrigation groups for lesion size, and pairwise comparisons were made with the Dwass-Steel-Critchlow-Fligner test. Before and after comparisons within each group, the Wilcoxon rank test was used. The significance level for the statistical analysis was set to p<0.05.

Additionally, intraobserver reliability was evaluated for fractal and lesion size measurements via the concordance correlation coefficient (CCC).

ELIGIBILITY:
Inclusion Criteria: Patients aged 18 years and over

* Patients who approved the Endodontic Consent Form and Study Participation Form
* Vertucci Class 1 single-rooted mandibular premolars with PAI score of 3 and above, requiring primary endodontic treatment with a diagnosis of apical periodontitis
* Vertucci Class 1 single-rooted mandibular premolars with PAI score of 3 and above, requiring retreatment with a diagnosis of apical periodontitis
* Patients with good oral hygiene

Exclusion Criteria: Patients with systemic diseases

* Immunosuppressive patients
* Pregnant patients
* Those with mobility of 2 and above,
* Those with periodontal pocket depth of 5 mm and above.
* Those with internal and external resorption,
* Those with teeth with vertical and horizontal root fractures

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-07-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Recep Tayyip Erdoğan University Faculty of Dentistry Department of Endodontics, Rize, Rize Province, Turkey (Türkiye)

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of 150 patients aged 18 years and over, a total of 18 patients who refused to participate or did not meet the inclusion criteria were excluded from the study, and 132 patients were included. 14 patients did not participate in the follow-up process. 118 patients were analyzed.
Groups:
- Group 5 (SWEEPS): A Fotona Er:YAG laser device (SWEEPS 600, Fotona) with an 8.5 mm long and 600 µm diameter tapered fiber tip was used for activation. The device was set to AutoSWEEPS mode with two ultrashort micropulses (25 μs) continuously changing at 0.3 W, 20 mJ, and 15 Hz. The tip was placed in the pulp chamber, and the solution was activated with the air and water settings turned off.
  root canal treatment and irrigation activation: After the teeth were isolated with a rubber dam, the endodontic access cavity was opened. Then, #10-15 K-type hand files were inserted into the canals, and after determining point 0.0 with the electronic apex locator, the working length was determined to be 0.5 mm shorter than this point and confirmed radiographically. When a discrepancy was observed, the apex locator was considered correct. The root canals were prepared with ProTaper Next up to 3 sizes larger than the initial diameter via a torque-controlled endodontic motor in 300 rpm/2-5.2 Ncm rotation mode. Between each file, the canals were irrigated with 5 ml of 2.5% NaOCl. In retreatment cases, after opening the access cavity under rubber dam isolation, the guta percha was removed with RT files, and the rest of the procedure was performed in the same manner as for primary root canal treatment.
Period: Overall Study
Arm/Group | Group 1 (MDA) | Group 2 (Sonic Activation) | Group 3 (PUI) | Group 4 (PIPS) | Group 5 (SWEEPS) | Control Group (Conventional Syringe Irrigation)
Started | 22 | 22 | 22 | 22 | 22 | 22
Completed | 22 | 18 | 22 | 19 | 20 | 17
Not Completed | 0 | 4 | 0 | 3 | 2 | 5
Not completed — Lost to Follow-up | 0 | 4 | 0 | 3 | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group (Conventional Syringe Irrigation) | Group 1 (MDA) | Group 2 (Sonic Activation) | Group 3 (PUI) | Group 4 (PIPS) | Group 5 (SWEEPS) | Total
Number analyzed (Participants) | 17 | 22 | 18 | 22 | 19 | 20 | 118
Age, Continuous [Mean (Full Range); unit: Years] | 53.2 [25 to 71] | 44.0 [18 to 73] | 48.8 [20 to 70] | 44.7 [21 to 65] | 43.2 [19 to 63] | 44.8 [26 to 74] | 46.2 [18 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 7 | 4 | 11 | 10 | 12 | 55
  Male | 6 | 15 | 14 | 11 | 9 | 8 | 63
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Pre-operative lesion diameter [Mean (Standard Deviation); unit: mm2] | 3.01 (1.21) | 2.79 (1.67) | 3.11 (1.42) | 3.17 (2.04) | 2.96 (1.28) | 2.43 (0.94) | 2.91 (1.42)
Pre-operative PAI score [Mean (Standard Deviation); unit: scores on a scale] — Periapical status is evaluated radiographically using the Periapical Index (PAI), which scores lesions from 1 to 5 according to increasing radiographic appearance, helps to achieve consensus among dropping in categorizing lesions: PAI 1-normal periapical structure; PAI 2-minor bone changes; PAI 3-bone changes with mineral loss; PAI 4-well-defined radiolucency; PAI 5-radiolucency with marked bone destruction. PAIs 1-2 categorized healed status, while 3-5 categorized unhealed. For each activation group, the mean PAI of participants was recorded as the group's PAI value in the data table.
  scores on a scale | 4.412 (0.507) | 4.136 (0.834) | 4.056 (0.802) | 4.318 (0.568) | 4.211 (0.787) | 4.100 (0.641) | 4.205 (0.689)
Pre-operative fractal dimension [Mean (Standard Deviation); unit: unitless] — Lesion healing after root canal treatment was objectively assessed using fractal analysis to quantify bone recovery and trabecular remodeling. Fractal analysis was performed on panoramic radiographs with the box-counting method. A standardized 30×30 pixel region of interest (ROI) was placed 1 mm apical to the root apex. Images were processed in ImageJ through 8-bit conversion, Gaussian filtering, subtraction, thresholding, binarization, erosion-dilation, inversion, skeletonization, and fractal dimension calculation.
  unitless | 1.216 (0.044) | 1.23 (0.04) | 1.25 (0.034) | 1.235 (0.049) | 1.249 (0.042) | 1.216 (0.025) | 1.232 (0.039)

OUTCOME MEASURES:

1. Primary Outcome: Post-operative Diameter of the Periapical Lesion
Description: Post-endodontic treatment, a reduction in the diameter of the periapical lesion may be observed, or the lesion may exhibit complete radiographic resolution. the largest dimension obtained was recorded as the preoperative lesion diameter
Time Frame: 1 year from completion of treatment to follow-up
Measure: Mean (Standard Deviation); unit: Post-operative lesion diameter- mm2
Arm/Group | Control Group (Conventional Syringe Irrigation) | Group 1 (MDA) | Group 2 (Sonic Activation) | Group 3 (PUI) | Group 4 (PIPS) | Group 5 (SWEEPS)
Number analyzed (Participants) | 17 | 22 | 18 | 22 | 19 | 20
Post-operative lesion diameter- mm2 | 2.07 (2.28) | 0.98 (1.65) | 1.12 (1.84) | 0.78 (1.58) | 0.33 (0.24) | 0.43 (0.64)

2. Other Pre Specified Outcome: Post-operative Fractal Dimension
Description: According to research, a high fractal dimension value indicates a more complex structure with fewer spaces between trabeculae, whereas a low fractal dimension value reflects a simpler structure with larger inter-trabecular spaces. The healing processes of lesions following root canal treatment can be objectively analyzed using the fractal analysis method, allowing for a quantitative evaluation of the degree of bone tissue healing and the remodeling of the trabecular architecture post-treatment.Fractal analysis (FA) was performed by an experienced oral and maxillofacial radiologist who was blinded to the activation method and used the fractal box counting method on panoramic radiographs. Images were processed in ImageJ through 8-bit conversion, Gaussian filtering, subtraction, thresholding, binarization, erosion-dilation, inversion, skeletonization, and fractal dimension calculation.
Time Frame: 1 year from completion of treatment to follow-up
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | Control Group (Conventional Syringe Irrigation) | Group 1 (MDA) | Group 2 (Sonic Activation) | Group 3 (PUI) | Group 4 (PIPS) | Group 5 (SWEEPS)
Number analyzed (Participants) | 17 | 22 | 18 | 22 | 19 | 20
unitless | 1.326 (0.046) | 1.338 (0.035) | 1.345 (0.025) | 1.311 (0.055) | 1.322 (0.038) | 1.3 (0.057)

3. Secondary Outcome: Post-operative Periapical Index (PAI) Score
Description: Periapical status is evaluated radiographically using the Periapical Index (PAI), which scores lesions from 1 to 5 according to increasing radiographic appearance, helps to achieve consensus among dropping in categorizing lesions. In most studies utilizing the PAI, scores of 1 and 2 are classified as 'successful' or 'healed,' whereas scores of 3, 4, and 5 are categorized as 'unsuccessful' or 'non-healed.' Classifying PAI scores <3 as healed and ≥3 as non-healed may facilitate communication between studies and the comparison of outcomes, particularly in follow-up studies; however, this approach may not provide detailed information regarding the progression of the disease. Lesion sizes on panoramic X-ray were classified according to the PAI classification. For each activation group, the mean PAI of participants was recorded as the group's PAI value in the data table.
Time Frame: 1 year from completion of treatment to follow-up
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Control Group (Conventional Syringe Irrigation) | Group 1 (MDA) | Group 2 (Sonic Activation) | Group 3 (PUI) | Group 4 (PIPS) | Group 5 (SWEEPS)
Number analyzed (Participants) | 17 | 22 | 18 | 22 | 19 | 20
scores on a scale | 2.647 (1.272) | 2.000 (0.976) | 1.778 (1.215) | 1.864 (0.941) | 1.421 (0.507) | 1.400 (0.754)

ADVERSE EVENTS:
Time Frame: up to 1 year after treatment
Arm/Group | Control Group (Conventional Syringe Irrigation) | Group 1 (MDA) | Group 2 (Sonic Activation) | Group 3 (PUI) | Group 4 (PIPS) | Group 5 (SWEEPS)
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22 | 0/22 | 0/22 | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 0/22 | 0/22 | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 0/22 | 0/22 | 0/22 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-06-30): https://cdn.clinicaltrials.gov/large-docs/03/NCT06991803/Prot_SAP_ICF_003.pdf